CLINICAL TRIAL: NCT06563011
Title: The Assessment of Nutritional Status of Patients With IPF and The Effectiveness of Nutritional Support
Brief Title: The Assessment of Nutritional Status of Patients With IPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: İrem Çağla Özel (Other)
Responsible Party: Sponsor-Investigator, İrem Çağla Özel, Principal Investigator, Ankara University
Organization: Ankara University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: İ06-370-23
Record Dates: First submitted 2024-08-09; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: idiopathic pulmonary fibrosis; nutritional assessment; dietary counselling
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dependent Sample (Other): Before-after measurements will be made in the dependent sample.
  Interventions: Other: Counselling

INTERVENTIONS:
Other: Counselling — Tailored Dietary Counselling

SUMMARY:
The aim of this study is to comprehensively evaluate the nutritional status of IPF patients and to evaluate the effectiveness of 3-month dietary counselling. In this study, the nutritional status of IPF patients followed in Atatürk Sanatorium Training and Research Hospital were comprehensively evaluated.

A comprehensive assessment were performed, including nutritional status, anthropometric measurements, body composition, hand dynamometer, pulmonary function, and food frequency. Also quality of life were assessed by SGRQ. Tailored dietary counselling were given to the patients and, patients were assessed at the end of the 3-month follow-up period in terms of same parameters.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is an irreversible interstitial lung disease of unknown etiology, characterized by progressive loss of lung function. IPF is a disease of advanced age. Preliminary studies of IPF indicate that nutritional status may affect quality of life and prognosis, but the clinical significance of nutritional status has not been investigated. Weight loss is recognized as a common complication of IPF. There is no study that comprehensively evaluates the nutritional status of IPF patients in Turkey. The aim of this study is to comprehensively evaluate the nutritional status of IPF patients and to evaluate the effectiveness of 3-month dietary counselling. In this study, the nutritional status of IPF patients followed in Atatürk Sanatorium Training and Research Hospital were comprehensively evaluated. A comprehensive assessment were performed, including nutritional status, anthropometric measurements, body composition, dynamometer, pulmonary function, and several questionnaires. so quality of life were assessed by SGRQ. All measurements were taken at the baseline. Then, tailored dietary counselling were given to the patients and, patients were assessed at the end of the 3-month follow-up period in terms of same parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with IPF

Exclusion Criteria:

* Not giving written consent

Ages: 60 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
The Effectiveness of Tailored Dietary Counselling in Patients with IPF on Pulmonary Function | 12 weeks
  The effect of dietary counselling on change from baseline in FVC values at 12 weeks were assessed.
The Effectiveness of Tailored Dietary Counselling in Patients with IPF on Pulmonary Function-2 | 12 weeks
  The effect of dietary counselling on change from baseline in DLCO values at 12 weeks were assessed.
The Effectiveness of Tailored Dietary Counselling in Patients with IPF on BMI | 12 weeks
  The effect of dietary counselling on change from baseline in BMI (kg/m2) at 12 weeks were assessed.
The Effectiveness of Tailored Dietary Counselling in Patients with IPF on Body Composition | 12 weeks
  The effect of dietary counselling on change from baseline in body composition measured by BIA at 12 weeks were assessed.
The Effectiveness of Tailored Dietary Counselling in Patients with IPF on Energy Intake | 12 weeks
  The effect of dietary counselling on change from baseline in energy intake (kcal/day) at 12 weeks were assessed.
The Effectiveness of Tailored Dietary Counselling in Patients with IPF on Dietary Intake | 12 weeks
  The effect of dietary counselling on change from baseline in carbohydrate, protein and fat intake (kcal/day) at 12 weeks were assessed.
The Effectiveness of Tailored Dietary Counselling in Patients with IPF on HRQL | 12 weeks
  The effect of dietary counselling on change from baseline in St. George Respiratory Questionnaire (SGRQ) score at 12 weeks were assessed. Scores range from 0-100. While score of zero indicates normal, and a score of 100 indicates impaired quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nurcan Yabancı Ayhan, PhD, Study Director — Ankara University
Locations (1):
- Atatürk Sanatorium Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Faverio P, Bocchino M, Caminati A, Fumagalli A, Gasbarra M, Iovino P, Petruzzi A, Scalfi L, Sebastiani A, Stanziola AA, Sanduzzi A. Nutrition in Patients with Idiopathic Pulmonary Fibrosis: Critical Issues Analysis and Future Research Directions. Nutrients. 2020 Apr 17;12(4):1131. doi: 10.3390/nu12041131. PMID 32316662